CLINICAL TRIAL: NCT05615142
Title: Phase I Study of Low Dose Radiotherapy and Concurrent SBRT in Combination With PD-1 Inhibitors in Advanced Non-small Cell Lung Cancer (NSCLC) .
Brief Title: Safety and Tolerability of Low Dose Radiotherapy Concurrent SBRT and PD-1 Inhibitors in Advanced NSCLC.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, You Lu, Chair of Department of Thoracic Cancer, Sichuan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ECLIPSE-01
Record Dates: First submitted 2022-11-02; First posted 2022-11-14 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: NSCLC; Low Dose Radiotherapy; Stereotactic Body Radiotherapy; PD-1 Inhibitor
MeSH Terms: interventions — Radiotherapy; Radiosurgery; Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LDRT+SBRT Combined with PD-1 Inhibitors (Experimental): Dose escalation cohort. DOSE LEVEL: Low Dose Radiotherapy (LDRT) dose from 2 Gy to 6Gy (2 Gy/f) + partial stereotactic body radiation therapy (SBRT) dose at 10 Gy to 30 Gy (10 Gy/f) + PD-1 inhibitor (dose as recommended in the instruction manual).
  Interventions: Radiation: Low Dose Radiotherapy; Radiation: stereotactic body radiation therapy; Drug: PD-1 Inhibitors

INTERVENTIONS:
Radiation: Low Dose Radiotherapy — LDRT at dose escalation levels: 2 Gy/1f, 4 Gy/2f, 6 Gy/3f with conventional external beam radiation.
  Other Names: LDRT
Radiation: stereotactic body radiation therapy — Partial SBRT at dose escalation levels: 10 Gy/1f, 20 Gy/2f, 30 Gy/3f.
  Other Names: SBRT
Drug: PD-1 Inhibitors — Patients will receive treatment with PD-1 inhibitor (dose as recommended in the instruction manual) every 3 weeks for a maximum of 48 months.

SUMMARY:
This pilot phase I trial aims to investigate the safety and tolerability of low dose radiotherapy (LDRT) and concurrent partial stereotactic body radiation therapy (SBRT) in combination with programmed cell death-1 (PD-1) inhibitors in Stage IV non-small cell lung cancer (NSCLC) patients who have failed standard therapy. At least 9 participants will be enrolled in this study. All will take part at West China Hospital, Sichuan University.

DETAILED DESCRIPTION:
This exploratory phase I study will be conducted in West China Hospital, Sichuan University. A dose escalation of low dose radiotherapy (LDRT) and partial SBRT, 3 patients per cohort (a total of 9 patients) will be enrolled to determine the maximum tolerated dose (MTD) and dose-limiting toxicity (DLT).

All eligible patients will receive LDRT + partial SBRT at different dose levels (decried as below), followed by PD-1 inhibitors starting within 7 days after radiation completed. PD-1 inhibitors will be given at doses as recommended in the instruction manual every 3 weeks until disease progression, unacceptable toxicities, the patient withdraws informed consent, or PD-1 inhibitors reaches a maximum of up to 48 months.

Patients in the dose escalation will receive LDRT + partial SBRT at 3 cohorts with increasing dose levels: 2 Gy (2 Gy/f) + 10 Gy (10 Gy/f) in 1 fraction in dose level 1; 4 Gy (2 Gy/f) + 20 Gy (10 Gy/f) in 2 fractions in dose level 2; 6 Gy (2 Gy/f) + 30 Gy (10 Gy/f) in 3 fractions in dose level 3.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent/assent for the trial.
2. Be ≥18 years of age on day of signing informed consent.
3. Patients with histologically or cytologically confirmed stage IV NSCLC.
4. Be willing to undergo repeat biopsy of tumor lesions according to the study protocol.
5. Patients who have failed the standard therapy, or who are unsuitable for standard treatment, or refuse chemotherapy.
6. At least one measurable lesion according to RECIST 1.1. A lesion that has previously received radiotherapy can be considered a target lesion only if this lesion is clearly progressed after radiotherapy.
7. The target lesions (irradiated lesions) are > 5cm in in diameter
8. ECOG 0-2.
9. Life expectancy of > 3 months.
10. Patients must have normal organ and bone marrow function as defined below: Total bilirubin </= 1.5 x upper limit of normal (ULN). Aminotransferase (AST) Serum Glutamic Oxaloacetic Transaminase (SGOT)/ Alanine Aminotransferase (ALT) Serum Glutamic-Pyruvic Transaminase (SGPT) <2.5 X institutional upper limit of normal (</= 5 X institutional ULN for subjects with liver metastases) *WBC >/= 3500/uL, ANC >/= 1500/uL *Platelets >/= 90K/ul *Hemoglobin >/= 9g/dL *Creatinine </= 1.5 x ULN, or creatinine clearance ≥ 50 ml/min（Cockcroft-Gault equation）. Coagulation: International Normalized Ratio (INR)≤ 1.5 × ULN, Partial thromboplastin time (PTT) ≤1.5 × ULN; left ventricular ejection fraction (LVEF) >/= 50% and QTcF (Fridericia's formula) ≤ 450ms
11. Patients has recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.
12. Wash out period for chemotherapy is more than ≥ 4 weeks, for targeted small molecule therapy ≥ 5 half-lives; palliative radiotherapy must have been completed for at least ≥ 2 weeks, chest radiotherapy must have been completed for at least ≥ 4 weeks, and major surgery must have been completed for ≥ 4 weeks.
13. Subjects with no severe pulmonary ventilation dysfunction, no acute heart failure, and no contraindication to radiotherapy as judged by the radiotherapist. Subjects who agree to receive immunotherapy and radiotherapy treatment.
14. Subjects should agree to use an adequate method of contraception.

Exclusion Criteria:

1. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis and/or spinal cord compression, etc.
2. With oncologic emergencies that require immediate treatment
3. EGFR/ALK/ROS-1 mutation or mutation status unknown.
4. Has evidence of interstitial lung disease or active and/or non-infectious pneumonitis (drug-induced pneumonia, radiation-induced pneumonia, etc.) requiring steroid therapy.
5. History of pulmonary fibrosis, pulmonary hypertension, severe irreversible airway obstruction disease
6. Patients with peripheral neuropathy.
7. Significant heart disease or impairment of cardiac function
8. Fluid accumulating in the third space, such as pericardial effusion, pleural effusion and peritoneal effusion that remains uncontrolled by aspiration or other treatment
9. Known allergy to drugs or excipients, known severe allergic reaction to any of the PD-1 monoclonal antibodies
10. Severe infection within 4 weeks prior to the start of study treatment, including but not limited to hospitalization for infection, bacteremia, or severe pneumonia; treatment with oral or intravenous antibiotics within 2 weeks prior to the start of study treatment; patients receiving prophylactic antibiotic therapy (e.g., to prevent urinary tract infection or exacerbation of COPD) are eligible for this study.
11. Known or suspected active autoimmune disease (congenital or acquired) such as uveitis, enterocolitis, hepatitis, pituitary inflammation, vasculitis, nephritis, thyroiditis, etc. (patients with vitiligo, or resolved childhood asthma may be enrolled; patients with type I diabetes with good insulin control may also be enrolled)
12. Known allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse Events and/or Dose Limiting Toxicities as a Measurement of Safety and Tolerability of Low Dose Radiotherapy, Concurrent SBRT and PD-1 Inhibitors in Advanced NSCLC. | 48 months

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | up to 48 months after the enrollment
  Investigator assessed PFS according to RECIST v1.1. Progression free survival is defined as time of enrollment to first evidence of progressive disease.
Overall Survival (OS) | up to 48 months after the enrollment
  OS is defined as the difference (in months) between the date of study enrollment to the date death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: You Lu, MD, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sharma P, Allison JP. The future of immune checkpoint therapy. Science. 2015 Apr 3;348(6230):56-61. doi: 10.1126/science.aaa8172. PMID 25838373
- [Background] Demaria S, Coleman CN, Formenti SC. Radiotherapy: Changing the Game in Immunotherapy. Trends Cancer. 2016 Jun;2(6):286-294. doi: 10.1016/j.trecan.2016.05.002. PMID 27774519
- [Background] Bernstein MB, Krishnan S, Hodge JW, Chang JY. Immunotherapy and stereotactic ablative radiotherapy (ISABR): a curative approach? Nat Rev Clin Oncol. 2016 Aug;13(8):516-24. doi: 10.1038/nrclinonc.2016.30. Epub 2016 Mar 8. PMID 26951040
- [Background] Bezjak A, Paulus R, Gaspar LE, Timmerman RD, Straube WL, Ryan WF, Garces YI, Pu AT, Singh AK, Videtic GM, McGarry RC, Iyengar P, Pantarotto JR, Urbanic JJ, Sun AY, Daly ME, Grills IS, Sperduto P, Normolle DP, Bradley JD, Choy H. Safety and Efficacy of a Five-Fraction Stereotactic Body Radiotherapy Schedule for Centrally Located Non-Small-Cell Lung Cancer: NRG Oncology/RTOG 0813 Trial. J Clin Oncol. 2019 May 20;37(15):1316-1325. doi: 10.1200/JCO.18.00622. Epub 2019 Apr 3. PMID 30943123
- [Background] Klug F, Prakash H, Huber PE, Seibel T, Bender N, Halama N, Pfirschke C, Voss RH, Timke C, Umansky L, Klapproth K, Schakel K, Garbi N, Jager D, Weitz J, Schmitz-Winnenthal H, Hammerling GJ, Beckhove P. Low-dose irradiation programs macrophage differentiation to an iNOS(+)/M1 phenotype that orchestrates effective T cell immunotherapy. Cancer Cell. 2013 Nov 11;24(5):589-602. doi: 10.1016/j.ccr.2013.09.014. Epub 2013 Oct 24. PMID 24209604
- [Background] Theelen WSME, Peulen HMU, Lalezari F, van der Noort V, de Vries JF, Aerts JGJV, Dumoulin DW, Bahce I, Niemeijer AN, de Langen AJ, Monkhorst K, Baas P. Effect of Pembrolizumab After Stereotactic Body Radiotherapy vs Pembrolizumab Alone on Tumor Response in Patients With Advanced Non-Small Cell Lung Cancer: Results of the PEMBRO-RT Phase 2 Randomized Clinical Trial. JAMA Oncol. 2019 Sep 1;5(9):1276-1282. doi: 10.1001/jamaoncol.2019.1478. PMID 31294749
- [Background] Herrera FG, Ronet C, Ochoa de Olza M, Barras D, Crespo I, Andreatta M, Corria-Osorio J, Spill A, Benedetti F, Genolet R, Orcurto A, Imbimbo M, Ghisoni E, Navarro Rodrigo B, Berthold DR, Sarivalasis A, Zaman K, Duran R, Dromain C, Prior J, Schaefer N, Bourhis J, Dimopoulou G, Tsourti Z, Messemaker M, Smith T, Warren SE, Foukas P, Rusakiewicz S, Pittet MJ, Zimmermann S, Sempoux C, Dafni U, Harari A, Kandalaft LE, Carmona SJ, Dangaj Laniti D, Irving M, Coukos G. Low-Dose Radiotherapy Reverses Tumor Immune Desertification and Resistance to Immunotherapy. Cancer Discov. 2022 Jan;12(1):108-133. doi: 10.1158/2159-8290.CD-21-0003. Epub 2021 Sep 3. PMID 34479871